CLINICAL TRIAL: NCT05637866
Title: Effect of Soy Milk for Cow's Milk on Intermediate Cardiometabolic Outcomes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials
Brief Title: SRMA of the Effect of Soy Milk vs Cow's Milk on Cardiometabolic Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CIHR - Soy vs cow's milk
Record Dates: First submitted 2022-11-10; First posted 2022-12-05 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Lipid Disorder; Metabolic Disease; Non-Alcoholic Fatty Liver Disease
Keywords: Cholesterol; triglycerides; apolipoprotein B; hemoglobin A1c; fasting plasma glucose; fasting plasma insulin; 2hr plasma glucose; body weight; body mass index; body fat; waist circumference; blood pressure; adiposity; fatty liver; NAFLD; CRP; Inflammation; HDL-C; LDL-C; Non-HDL-c; Intrahepatocellular lipids; ALT; AST
MeSH Terms: conditions — Cardiovascular Diseases; Lipid Metabolism Disorders; Metabolic Diseases; Non-alcoholic Fatty Liver Disease; Body Weight; Obesity; Fatty Liver; Inflammation | interventions — Soy Milk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Soy Milk: Soy milk beverage
  Interventions: Other: Soy milk

INTERVENTIONS:
Other: Soy milk — Soya milk or soymilk, a plant-based beverage that can be sweetened or unsweetened.

SUMMARY:
Dairy consumption has shown associations with decreased incidence of cardiometabolic diseases. With the growing interest in plant-based eating, and the mounting evidence for the cardiovascular benefits of plant forward diets, national dietary guidelines have pivoted away from promoting exclusive daily dairy consumption. Soymilk is the most nutritionally comparable non-dairy plant-based alternative to cow's milk. Although the DGA, Health Canada, and various pediatric associations recognize fortified soymilk as the only non-dairy alternative equivalent to cow's milk and it can carry an approved health claim for coronary heart disease risk reduction based on the soy protein that it contains, soymilk is classified by the NOVA classification as an ultra-processed food (the opposite of the classification of cow's milk as an unprocessed or minimally processed food). To be an acceptable iso-sweet alternative to cow's milk, soymilk is also often sweetened with sucrose, which is designated as an added sugar, whereas the lactose that sweetens cow's milk is not (despite lactose in cow's milk being present in quantities that are double that of sucrose in soymilk products designed to be iso-sweet analogues of cow's milk). With near universal recommendations from major public health authorities to reduce the intake of both ultra-processed foods and added sugars and the FDA proposing to update its "healthy" claim criteria to limit added sugars, the role of soymilk as a "healthy" non-dairy alternative to cow's milk is in serious question. The effect of soy protein on other cardiometabolic outcomes is also unclear. To address this question and better inform health claims and guideline development, the investigators will conduct a systematic review and meta-analysis of randomized controlled trials of the effect of soy protein as soy milk, in substitution for cow's milk, on various intermediate cardiometabolic mediators.

DETAILED DESCRIPTION:
RATIONALE. Soymilk and other processed soy products are at an important crossroads. Although the DGA, Health Canada, and various pediatric associations recognize fortified soymilk as the only non-dairy plant milk alternative equivalent to cow's milk and it can carry an approved health claim for coronary heart disease risk reduction based on the soy protein that it contains, soymilk is classified by the NOVA classification as an ultra-processed food (the opposite of the classification of cow's milk as an unprocessed or minimally processed food). To be an acceptable iso-sweet alternative to cow's milk, soymilk is also often sweetened with sucrose, which is designated as an added sugar, whereas the lactose that sweetens cow's milk is not (despite lactose in cow's milk being present in quantities that are double that of sucrose in soymilk products designed to be iso-sweet analogues of cow's milk). With near universal recommendations from major public health authorities to reduce the intake of both ultra-processed foods and added sugars and the FDA updating its "healthy" claim criteria to limit added sugars, the role of soymilk as a "healthy" non-dairy alternative to cow's milk is in serious question.

OBJECTIVES. The objective is to conduct a systematic review and meta-analysis of randomized controlled trials to assess the effect of soymilk in substitution for cow's milk and its modification by added sugars (sweetened versus unsweetened) on established cardiometabolic risk factors of clinical and public health importance and assess the certainty of the evidence using the Grading of Recommendations Assessment Development and Evaluation (GRADE) system.

DESIGN. The systematic review and meta-analyses will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting items for Systematic Reviews and Meta-Analyses (PRISMA).

DATA SOURCES. Medline, Embase, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by manual searches of references of included studies.

STUDY SELECTION. Randomized controlled trials of ≥3-weeks assessing the effect of soy milk in substitution for cow's milk on cardiometabolic risk factors will be included.

DATA EXTRACTION. Two or more investigators will independently extract relevant data. Authors will be contacted for additional information and any missing data will be computed/imputed using standard formulae.

RISK OF BIAS. Two or more investigators will independently assess risk of bias using the Cochrane Risk of Bias Tool 2. All disagreements will be resolved by consensus.

OUTCOMES. Outcomes will include changes in established markers of (1) adiposity (body weight, BMI, body fat, waist circumference, abdominal fat); (2) glycemic control (HbA1c, fasting plasma glucose (FPG), fasting plasma insulin (FPI), plasma glucose area under the curve (AUC), and 2h plasma glucose (2hPG)); (3) blood lipids (LDL-cholesterol, non-HDL-cholesterol, apolipoprotein B, HDL-cholesterol, triglycerides); (4) blood pressure (systolic blood pressure and diastolic blood pressure); (5) non-alcoholic fatty liver disease (NAFLD) (intrahepatocellular lipids (IHCL), alanine transaminase (ALT), aspartate aminotransferase (AST), and fatty liver index (FLI)); (6) inflammation (C-reactive protein (CRP)); (7) renal function and structure (creatinine, creatinine clearance (CrCl), glomerular filtration rate (GFR), estimated GFR (eGFR), albuminuria, albumin-to-creatinine ratio (ACR)); and (8) and uric acid.

DATA SYNTHESIS. Data will be pooled using the Generic Inverse Variance method for each outcome. As one of our primary research questions relates to the role of added sugars as a mediator in any observed differences between soy milk and cow's milk, we will stratify results by the presence of added sugars in soy milk (sweetened versus unsweetened) and assess effect modification by this variable on pooled estimates. Random effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover design trials. Heterogeneity will be assessed (Cochran Q statistic) and quantified (I2 statistic). Sources of heterogeneity will be explored (if there are >=10 trial comparisons) by sensitivity analyses and a priori subgroup analyses (dose, comparator, follow-up, baseline levels, design, age, health status, funding and risk of bias). Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. Publication bias will be assessed (if there are >=10 trial comparisons) by inspection of funnel plots and the Egger and Begg tests. Adjustment for evidence of funnel plot asymmetry or small study effects will be conducted by the Duval and Tweedie trim-and-fill method.

GRADE ASSESSMENT. To assess the certainty of the evidence, the investigators will use the GRADE system, an evidence-based grading system adopted by >100 organizations (http://www.gradeworkinggroup.org/). It grades the evidence as high, moderate, low or very low quality based on the study design and a series of downgrades (risk of bias, imprecision, inconsistency, indirectness, publication bias) and upgrades (large magnitude of the effect, dose-response gradient, and attenuation by confounding). The investigators will follow the GRADE handbook (https://gdt.gradepro.org/app/handbook/ handbook.html) and use the GRADEpro GDT (gradepro.org) software.

ADD-ON SYNTHESIS (LACTOSE VERSUS ADDED SUGARS) To interrogate the question of the role of added sugars as a mediator of any observed effects of sweetened soymilk, we will conduct a sub-synthesis (a separate systematic review and meta-analysis of RCTs) of the effect of lactose (which is not considered an added sugar) versus added sugars (sucrose, HFCS, or fructose) irrespective of matrix (all comparisons with a matched matrix will be included). We will follow the same protocol and analysis plan as that for the main analysis.

KNOWLEDGE TRANSLATION PLAN. The investigators will follow the Ottawa model of Research for knowledge translation. The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact journals. Target audiences will include public health and clinical communities with an interest in nutrition and cardiometabolic diseases. Feedback will be incorporated and used to improve public health messages and key areas for future research will be defined. The PIs will network among opinion leaders to increase awareness and participate directly in the development of future guidelines.

SIGNIFICANCE. Both proposed projects will aid in knowledge translation related to the role of soy milk as a "healthy" non-dairy alternative to cow's milk, strengthening the evidence-base for guidelines development in the U.S., Canada, Europe, and beyond and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials
* Soy milk intervention
* Cow's milk comparator
* Intervention duration ≥ 3 weeks
* Data for at least 1 outcome

Exclusion Criteria:

* Non-human studies
* Observational studies
* Acute single-bolus feeding studies
* Participants < 18 years of age
* Multimodal interventions
* Lack of suitable comparator
* Intervention duration < 3 weeks
* No viable outcome data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with or without cardiovascular risk factors
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Blood lipids - LDL-Cholesterol (LDL-C) | Immediately after the intervention
  LDL-C mean difference and 95% CIs in mmol/L
Blood lipids - HDL-Cholesterol (HDL-C) | Immediately after the intervention
  HDL-C mean difference and 95% CIs in mmol/L
Blood lipids - Triglycerides (TG) | Immediately after the intervention
  TG mean difference and 95% CIs in mmol/L
Blood lipids - non-HDL-Cholesterol (Non HDL-C) | Immediately after the intervention
  Non-HDL-C mean difference and 95% CIs in mmol/L
Blood lipids - Apolipoprotein B (ApoB) | Immediately after the intervention
  ApoB mean difference and 95% CIs in g/L
Glycemic control - Hemoglobin A1c (HbA1c) | Immediately after the intervention
  HbA1c mean difference and 95% CIs in %
Glycemic control - fasting plasma glucose (FPG) | Immediately after the intervention
  FPG mean difference and 95% CIs in mmol/L
Glycemic control - fasting plasma insulin (FPI) | Immediately after the intervention
  FPI mean difference and 95% CIs in mmol/L
Glycemic control - glucose tolerance - plasma glucose area under the curve (AUC) | Immediately after the intervention
  AUC mean difference and 95% CIs in mmol x min/l
Glycemic control - glucose tolerance - 2h plasma glucose (2h-PG) | Immediately after the intervention
  2h plasma glucose (2h-PG) during a 75g oral glucose tolerance test (OGTT) in mmol/L
Adiposity - Body weight | Immediately after the intervention
  Body weight mean difference and 95% CIs in kg
Adiposity - Body mass index (BMI) | Immediately after the intervention
  BMI mean difference and 95% CIs in kg/m2
Adiposity - Body fat | Immediately after the intervention
  Body fat mean difference and 95% CIs in %
Adiposity - Waist circumference | Immediately after the intervention
  Waist circumference mean difference and 95% CIs in cm
Blood pressure - systolic blood pressure (SBP) | Immediately after the intervention
  SBP mean difference and 95% CIs in mmHg
Blood pressure - diastolic blood pressure (DBP) | Immediately after the intervention
  DBP mean difference and 95% CIs in mmHg
Markers of non-alcoholic fatty liver disease (NAFLD) - Intrahepatocellular lipids (IHCL) | Up to 20 years
  IHCL mean difference and 95% CIs in %
Markers of non-alcoholic fatty liver disease (NAFLD) - alanine transaminase (ALT) | Immediately after the intervention
  ALT mean difference and 95% CIs in U/L
Markers of non-alcoholic fatty liver disease (NAFLD) - aspartate aminotransferase (AST) | Immediately after the intervention
  AST mean difference and 95% CIs in U/L
Markers of non-alcoholic fatty liver disease (NAFLD) - fatty liver index (FLI) | Immediately after the intervention
  FLI mean difference and 95% CIs
Markers of inflammation - C-reactive protein (CRP) | Immediately after the intervention
  CRP mean difference and 95% CIs in mg/dL
Renal function and structure - creatinine | Immediately after the intervention
  Creatinine mean difference and 95% CIs in mcmol/L
Renal function and structure - creatinine clearance (CrCl) | Immediately after the intervention
  CrCl mean difference and 95% CIs in mL/min
Renal function and structure - glomerular filtration rate (GFR) | Immediately after the intervention
  GFR mean difference and 95% CIs in ml/min/1.73 m2
Renal function and structure - estimated GFR (eGFR) | Immediately after the intervention
  eGFR mean difference and 95% CIs in ml/min/1.73 m2
Renal function and structure - albumin excretion rate (AER) | Immediately after the intervention
  AER mean difference and 95% CIs in mg/L
Renal function and structure - albumin-to-creatinine ratio (ACR) | Immediately after the intervention
  ACR mean difference and 95% CIs in mg/mmol creatinine
Uric acid | Immediately after the intervention
  Uric acid in mcmol/L

CONTACTS AND LOCATIONS:
Overall Officials: John L. Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no individual data collected. However, data from all included studies will be published in the manuscript and supplementary material

REFERENCES:
- [Background] Malik VS, Sun Q, van Dam RM, Rimm EB, Willett WC, Rosner B, Hu FB. Adolescent dairy product consumption and risk of type 2 diabetes in middle-aged women. Am J Clin Nutr. 2011 Sep;94(3):854-61. doi: 10.3945/ajcn.110.009621. Epub 2011 Jul 13. PMID 21753066
- [Background] Maersk M, Belza A, Stodkilde-Jorgensen H, Ringgaard S, Chabanova E, Thomsen H, Pedersen SB, Astrup A, Richelsen B. Sucrose-sweetened beverages increase fat storage in the liver, muscle, and visceral fat depot: a 6-mo randomized intervention study. Am J Clin Nutr. 2012 Feb;95(2):283-9. doi: 10.3945/ajcn.111.022533. Epub 2011 Dec 28. PMID 22205311
- [Background] McGregor RA, Poppitt SD. Milk protein for improved metabolic health: a review of the evidence. Nutr Metab (Lond). 2013 Jul 3;10(1):46. doi: 10.1186/1743-7075-10-46. PMID 23822206
- [Derived] Erlich MN, Ghidanac D, Blanco Mejia S, Khan TA, Chiavaroli L, Zurbau A, Ayoub-Charette S, Almneni A, Messina M, Leiter LA, Bazinet RP, Jenkins DJA, Kendall CWC, Sievenpiper JL. A systematic review and meta-analysis of randomized trials of substituting soymilk for cow's milk and intermediate cardiometabolic outcomes: understanding the impact of dairy alternatives in the transition to plant-based diets on cardiometabolic health. BMC Med. 2024 Aug 22;22(1):336. doi: 10.1186/s12916-024-03524-7. PMID 39169353
- See also: Canada's Food Guide — https://food-guide.canada.ca/en/healthy-eating-recommendations/